CLINICAL TRIAL: NCT01718418
Title: Prebiotics and Probiotics as Means to Modulate Colonic Events, With Specific Focus on Metabolism and Satiety
Brief Title: Role of Colonic Events on Metabolism and Appetite Control: A Synbiotic Approach
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Lund University (Other)
Responsible Party: Principal Investigator, Elin Johansson, MSc, post-graduate student, Lund University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: Dnr2010/457
Record Dates: First submitted 2012-10-09; First posted 2012-10-31 (Estimated); Last update posted 2013-05-08 (Estimated); Status verified 2013-05

CONDITIONS: Obesity; Metabolic Syndrome
MeSH Terms: conditions — Obesity; Metabolic Syndrome

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- + ind.CHO + prebiotics (Experimental): test meal: intrinsic indigestible carbohydrates in combination with a combined probiotic supplement.
  Interventions: Other: test meal
- + ind.CHO - prebiotics (Experimental): test meal: intrinsic indigestible carbohydrates in combination with placebo probiotic supplement.
  Interventions: Other: test meal
- - ind.CHO - prebiotics (Experimental): reference: no ind. carbohydrates and no probiotic supplement
  Interventions: Other: reference

INTERVENTIONS:
Other: test meal
  Arms: + ind.CHO + prebiotics; + ind.CHO - prebiotics
Other: reference
  Arms: - ind.CHO - prebiotics

SUMMARY:
The purpose of the study is to evaluate food factors related to colonically derived regulation of glucose metabolism (and related parameters) and satiety using a semi-acute meal study in healthy subjects as experimental model.

ELIGIBILITY:
Inclusion Criteria:

* Normal fasting blood glucose, BMI 19-25 kg/m2, for women: hormon based contraceptives

Exclusion Criteria:

* gastrointestinal diseases or food allergies e.g. lactose-, gluten intolerance, metabolic disorders e.g. diabetes, tobacco/snuff users. Antibiotic or probiotic usage within two weeks, and during the study. Vegetarians

Ages: 20 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 21 (Actual)
Dates: Start 2012-09; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Differences in concentration of risk markers in blood, measured post-prandial after a breakfast meal. | Post-prandially after breakfast, 0-210 min
  Variables (blood glucose, insulin, incretin, inflammatory markers, markers of colonic fermentation) are measured after two-weeks ingestion of test products. The experimental day is terminated after a lunch meal.

SECONDARY OUTCOMES:
voluntary energy intake | Post-prandially after breakfast, 0-210 min
  Energy intake at lunch is measured after two-weeks ingestion of test products. The experimental day is terminated after the lunch meal.
Subjective satiety | post-prandially after breakfast, 0-210 min
  The subjective sensation of satiety, hunger and desire to eat is measured using a (VAS) questionnaire.
Differences in gut microbiota | Faecal samples are collected after 14 days intake of test- and reference product
  The effect on gut microbiota of 14 days intake of test- and reference product are investigated in faecal samples.

CONTACTS AND LOCATIONS:
Overall Officials: Anne Nilsson, PhD, Principal Investigator — Lund University
Locations (1):
- Applied Nutrition and Food Chemistry, Lund University, Lund, Sweden

REFERENCES:
- [Derived] Nilsson A, Johansson-Boll E, Sandberg J, Bjorck I. Gut microbiota mediated benefits of barley kernel products on metabolism, gut hormones, and inflammatory markers as affected by co-ingestion of commercially available probiotics: a randomized controlled study in healthy subjects. Clin Nutr ESPEN. 2016 Oct;15:49-56. doi: 10.1016/j.clnesp.2016.06.006. Epub 2016 Jul 2. PMID 28531784